CLINICAL TRIAL: NCT01048502
Title: Fenofibrate and Omega-3 Fatty Acid Modulation of Endotoxemia: The FFAME Study
Brief Title: Fenofibrate and Omega-3 Fatty Acid Modulation of Endotoxemia
Acronym: FFAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 810598; P50HL083799 (NIH)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease
Keywords: healthy volunteer
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fenofibrate; Tablets; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fenofibrate (Tricor) (145 mg/day) (Experimental): Participants will be given 1 fenofibrate (Tricor) 145mg and 4 fish oil placebos - supplies of study drug will be provided to last 8 weeks.
  Interventions: Drug: Fenofibrate (Tricor) tablets
- Placebo (Placebo Comparator): Participants will be given 5 placebo pills (4 fish oil placebo and 1 fenofibrate placebo) - supplies of study drug will be provided to last 8 weeks.
  Interventions: Drug: Placebo
- Lovaza (900 mg/day) (Experimental): Participants will be given 1 Lovaza capsule, 3 Fish oil placebo capsules, and 1 Fenofibrate placebo - supplies of study drug will be provided to last 8 weeks.
  Interventions: Drug: Lovaza
- Lovaza (3,600 mg/day) (Experimental): Participants will be given 4 Lovaza capsules and 1 Fenofibrate placebo - supplies of study drug will be provided to last 8 weeks.
  Interventions: Drug: Lovaza

INTERVENTIONS:
Drug: Fenofibrate (Tricor) tablets — One 145 mg tablet taken once daily, in the evening, with food, for 6 to 8 weeks
  Arms: Fenofibrate (Tricor) (145 mg/day)
Drug: Placebo — Two placebo capsules taken twice daily, morning and evening, with food and one placebo gel capsule taken once daily, in the evening, with food, for 6 to 8 weeks
  Arms: Placebo
Drug: Lovaza — 900 mg/day: One 900 mg capsule taken once daily, morning or evening; or 3,600 mg/day: Two 900 mg capsules taken twice daily, morning and evening; All capsules to be taken with food, for 6 to 8 weeks.
  Arms: Lovaza (3,600 mg/day); Lovaza (900 mg/day)

SUMMARY:
The purpose of this study is to better understand the anti-inflammatory benefits of two prescription medicines that are currently used to help people with cholesterol problems.

Fish oil, from eating certain kinds of fish and from supplement pills, has been used to help control cholesterol and reduce inflammation (the body's response to injury or sickness). Lovaza® is the brand name for prescription strength fish oil pills. In this study, we will be looking at how Lovaza® works to help reduce inflammation in healthy volunteers.

Tricor® is the brand name for prescription fenofibrate pills. Fenofibrate is a prescription medicine that many doctors give to people with high triglyceride (fat in the blood) levels. In this study, we will be looking at how Tricor® works to help reduce inflammation in healthy volunteers.

Endotoxin or lipopolysaccharide (LPS) is a small part of bacteria (that is no longer living) that can cause many of the effects similar to bacterial infections in humans. However, it can be administered in very small amounts to produce a mild immune response much the same as a 'flu' like illness. Within 1 ½ -3 hours after giving LPS by vein, a response consisting of fever, chills, headache, nausea and vomiting and generalized aches and pains will occur which lasts up to 6-8 hours. In addition to the flu like symptoms, the response causes temporary changes in cholesterol, triglycerides and blood sugar. Different people respond differently to LPS. We are using LPS in this study to bring on a temporary inflammatory response in the body and to compare the responses of people who receive Lovaza® or Tricor® to the responses of people who receive a placebo (pill that does not contain medicine).

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant/lactating women between the ages of 18 and 45.
* Body Mass Index (BMI) ≥18 and ≤30
* Participants who are able to give written informed consent and willing to comply with all study-related procedures.

Exclusion Criteria:

* Known clinically manifest atherosclerotic cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease
* History of diabetes mellitus
* Fasting glucose >126mg/dL at screening
* History of a non-skin malignancy within the previous 5 years
* Renal insufficiency as defined by creatinine outside of lab defined normal range or eGFR <60 ml/Kg/min at Screening Visit
* History of liver disease or abnormal Liver Function Tests (LFTs) (aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase, gamma-glutamyl transpeptidase (GGT) > 1.5x upper limit of normal (ULN); bilirubin > 2x ULN) at Screening Visit
* Men who are unwilling to limit alcohol consumption to < 14 alcoholic drinks per week or < 4 alcoholic drinks per occasion (American Medical Association/National Institute on Alcohol Abuse and Alcoholism (AMA / NIAAA) criteria for "at risk" usage levels) while participating in the study
* Women who are unwilling to limit alcohol consumption to < 7 alcoholic drinks per week or < 3 alcoholic drinks per occasion (AMA / NIAAA criteria for "at risk" usage levels) while participating in the study
* Total white blood cell count less than or equal to 3.0 THO/uL
* Hemoglobin less than 11.0 g/dL
* Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition or minor active infection
* Self-reported history of HIV positive
* First degree family history of premature cardiovascular disease event (father or brother if diagnosed at before 55 years of age; mother or sister if diagnosed before 65 years of age)
* Patients who have undergone any organ transplant
* Individuals who currently use tobacco products or have done so in the previous 30 days
* Treatment with aspirin, Nonsteroidal Anti-inflammatory Drugs (NSAIDs), cyclooxygenase-2 (COX-2) inhibitors, steroids or any immunomodulatory therapy 2 weeks prior to the Screening Visit
* Treatment with statins, fibrates or niacin 4 weeks prior to the Screening Visit.
* Current daily use of Vitamin C > 1000 mg, Beta carotene > 1000 IU, vitamin A > 5000 IU, vitamin E > 400 IU, and selenium > 200 mcg
* Participants who are unwilling to eliminate omega-3 fatty acid (eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA)) supplements and/or fortified food, or have their usual intake of high omega-3 fish (tuna and other non-fried fish) be > 3 to 4 servings per month as assessed by a simple screening questionnaire
* Positive urine pregnancy test result.
* Participation in another clinical trial within the previous 6 weeks prior to the Screening Visit.
* Poorly controlled blood pressure (BP > 160/110) or on any anti-hypertensive medications.
* A diagnosis of metabolic syndrome using updated 2004 National Cholesterol Education Program Adult Treatment Panel III (NCEP ATPIII) criteria.
* Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muredach P Reilly, MB, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical and Translational Research Center (CTRC); Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ferguson JF, Xue C, Hu Y, Li M, Reilly MP. Adipose tissue RNASeq reveals novel gene-nutrient interactions following n-3 PUFA supplementation and evoked inflammation in humans. J Nutr Biochem. 2016 Apr;30:126-32. doi: 10.1016/j.jnutbio.2015.12.010. Epub 2016 Jan 11. PMID 27012629
- [Derived] Mulvey CK, Ferguson JF, Tabita-Martinez J, Kong S, Shah RY, Patel PN, Master SR, Usman MH, Propert KJ, Shah R, Mehta NN, Reilly MP. Peroxisome Proliferator-Activated Receptor-alpha Agonism With Fenofibrate Does Not Suppress Inflammatory Responses to Evoked Endotoxemia. J Am Heart Assoc. 2012 Aug;1(4):e002923. doi: 10.1161/JAHA.112.002923. Epub 2012 Aug 24. PMID 23130172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects were enrolled; 80 completed the study.
Period: Overall Study
Arm/Group | Fenofibrate (Tricor) (145 mg/Day) | Placebo | Lovaza (900 mg/Day) | Lovaza (3,600 mg/Day)
Started | 24 | 23 | 28 | 25
Completed | 20 | 16 | 23 | 21
Not Completed | 4 | 7 | 5 | 4
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 5 | 3
Not completed — Physician Decision | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fenofibrate (Tricor) (145 mg/Day): Participants will be given 1 fenofibrate (Tricor) 145mg and 4 fish oil placebos - supplies of study drug will be provided to last 8 weeks.
  Fenofibrate (Tricor)tablets: One 145 mg tablet taken once daily, in the evening, with food, for 6 to 8 weeks
- Total: Total of all reporting groups
Arm/Group | Fenofibrate (Tricor) (145 mg/Day) | Placebo | Lovaza (900 mg/Day) | Lovaza (3,600 mg/Day) | Total
Number analyzed (Participants) | 24 | 23 | 28 | 25 | 100
Age, Continuous [Mean (Full Range); unit: years] | 25.58 [21 to 43] | 25.96 [18 to 43] | 26.68 [18 to 42] | 24.68 [19 to 36] | 25.75 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 12 | 12 | 47
  Male | 13 | 11 | 16 | 13 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 3 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 8 | 5 | 22
  White | 16 | 14 | 17 | 16 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Omega-3 Fatty Acid Supplementation on Cytokine Production (Plasma Levels of TNFα) During an in Vivo Inflammatory Challenge (LPS).
Time Frame: randomization and 8 weeks post
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Lovaza (900 mg/Day) | Lovaza (3,600 mg/Day)
Number analyzed (Participants) | 16 | 23 | 21
pg/mL
  TNF-α at randomization | 0.95 [0.8 to 1.68] | 1.26 [0.72 to 1.76] | 1.14 [0.76 to 1.81]
  TNF-α 8 weeks post randomization | 1.12 [0.64 to 1.84] | 1.25 [0.78 to 1.76] | 0.99 [0.64 to 1.34]

2. Secondary Outcome: Changes in Inflammatory Parameter (Plasma TNF-α Levels) After Treatment With Fenofibrate or Placebo.
Time Frame: baseline and 6-8 weeks
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Fenofibrate (Tricor) (145 mg/Day) | Placebo
Number analyzed (Participants) | 20 | 16
pg/mL
  TNF-α at randomization | 1.2 (0.5) | 1.5 (1.2)
  TNF-α 6-8 weeks post randomization | 1.1 (0.4) | 0.2 (1.1)

ADVERSE EVENTS:
Groups:
- Tricor (145 mg/Day): Participants will be given 1 Tricor 145mg and 4 fish oil placebos - supplies of study drug will be provided to last 8 weeks.
  Fenofibrate tablets: One 145 mg tablet taken once daily, in the evening, with food, for 6 to 8 weeks
Arm/Group | Tricor (145 mg/Day) | Placebo | Lovaza (900 mg/Day) | Lovaza (3,600 mg/Day)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 4/24 | 3/23 | 8/28 | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tricor (145 mg/Day) (N=24) | Placebo (N=23) | Lovaza (900 mg/Day) (N=28) | Lovaza (3,600 mg/Day) (N=25)
> 2g drop in Hgb from baseline (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
cold/allergy symptoms (General disorders) | 3 (3) | 2 (2) | 4 (4) | 7 (7) — Subjects reported having illnesses that were unrelated to study but that occurred during participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes